CLINICAL TRIAL: NCT00456235
Title: Interruption of the Calcineurine Inhibitors (ICN) and Introduction of Mycophenolate Mofetil (MMF) in Liver Transplant Patients With Side Effects Due to ICN: Study of the Reduction of the Risks of Rejection by Mycophenolate Mofetil Therapeutic Drug Monitoring
Brief Title: Reduction in the Risk of Rejection by Mycophenolate Mofetil Dose Adjustment in Liver Transplant Patients With Side Effects Caused by the Calcineurine Inhibitors
Acronym: MONOCEPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I06024
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Tacrolimus

ARMS (2):
- adjument MMF (Experimental): adjusting the dose according to the MMF AUC of mycophenolic acid
  Interventions: Drug: Mycophénolate Mofétil; Drug: Ciclosporine A; Drug: Tacrolimus
- continued treatment (Active Comparator): Continued treatment empirically usual
  Interventions: Drug: Mycophénolate Mofétil; Drug: Ciclosporine A; Drug: Tacrolimus

INTERVENTIONS:
Drug: Mycophénolate Mofétil
Drug: Ciclosporine A
Drug: Tacrolimus

SUMMARY:
The aim of this project is to determine whether, in liver transplant patients with side effects due to ICN, the use of MMF in monotherapy can be optimised by dose adjustment based on the area under the curve (AUC) of mycophenolic acid (MPA). It involves a multicentre phase IV trial with direct individual benefit.

A population of 130 liver transplant patients at 2 to 10 years post-transplant, showing significant clinical ICN side effects and being given bitherapy by ICN +MMF will be included and randomised 1:1 in two arms:

* Arm 1: progressive interruption of ICN after obtaining an AUC of MPA of 50 mg.h/l, followed by MMF monotherapy with dose adjustment based on the AUC of MPA,
* Arm 2: continuation of the ICN+MMF bitherapy without MMF therapeutic drug monitoring.

The main judgement criterion will be the incidence of acute rejection in the 2 groups at 6 months. The secondary judgment criterion will be the evaluation of the benefit of stopping ICN on the side effects caused by these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patient with first liver transplantion or retransplantation since more than 6 months: with a post-transplant lapse of time of 2 to 10 years and showing one of the following adverse effects of ICN:
* Renal insufficiency defined by a creatinine clearance <50ml/mn (calculated or estimated according to the Cockcroft formula)
* Arterial hypertension not controlled by an anti-hypertensive bitherapy
* Diabetes mellitus (fasting glycaemia >7.0mmol/l), whether treated or not
* Neuromuscular toxicity
* Immunosuppression by cyclosporine or tacrolimus and MMF
* Hepatic biopsy performed within the 6 months preceding the inclusion for the patients with a post-transplant period of <5 years and in the 12 months preceding the inclusion for patients with a post transplant period of >5 years.

Exclusion Criteria:

* Acute rejection within the 6 months preceding the screening
* Previous history of cortico-resistant rejection
* Chronic rejection
* Significant ductopenia (absence of inter-lobule biliary canals in more than 30% of the portal tracts) on the pre-screening biopsy.
* Existence of a pre-transplantation diabetes mellitus.
* Liver transplantation for auto-immune hepatitis or primary sclerosing cholangitis
* Patients transplanted for viral C cirrhosis with reinfection lesions of the transplanted organ, rendering treatment by ribarivine + interferon conceivable in the year following inclusion.
* Counter-indications to MMF (anaemia, leucopenia)
* Immunosuppression by sirolimus, everolimus, azathioprine or corticoids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy proven acute rejection treated | 6 months
  Incidence of biopsy proven acute rejection treated with corticoids or requiring a re-introduction of ICN in arm 1 -- or an increase of ICN in arm 2 -- 6 months after the interruption of ICN (arm 1) or after randomization (arm 2).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MARQUET, MD, Principal Investigator — CHU Limoges
Locations (17):
- France (17):
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - Hôpital Edouard Herriot, Lyon
  - CHU de Marseille, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nice, Nice
  - Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - Hôpital Paul Brousse, Villejuif